CLINICAL TRIAL: NCT01463163
Title: Ticagrelor in Comparison to Prasugrel for Early Inhibition of Platelet Reactivity in Patients With ST-elevation Myocardial Infarction (STEMI), Undergoing Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-8
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Platelet Reactivity
Keywords: Platelet reactivity; Ticagrelor; Prasugrel
MeSH Terms: interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator): Prasugrel 60mg LD followed by 10mg MD starting post 24 hours
  Interventions: Drug: Prasugrel
- Ticagrelor (Experimental): Ticagrelor 180mg LD followed by 90mg x2 MD starting post 12±6 hours
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 60mg LD followed by 10mg x1 MD starting post 24 hours
  Arms: Prasugrel
Drug: Ticagrelor — Ticagrelor 180mg LD followed by 90mg x2 MD starting after 12±6 hours
  Arms: Ticagrelor

SUMMARY:
This is a single-center, randomized, single-blind, investigator-initiated, pharmacodynamic study with a parallel design. Patients with ST elevation myocardial infarction, undergoing primary percutaneous coronary intervention will be randomized after informed consent, in a 1:1 ratio to the following treatment groups:

Group Α: Ticagrelor 180mg loading dose (LD), followed by a 90mg x2 maintenance dose (MD)starting 12±6 hours post LD, until Day 5 (5 days after randomization) Group Β: Prasugrel 60 mg LD followed by 10mg x1 MD starting 24 hours post LD, until Day 5 (5 days after randomization).

Platelet reactivity assessment will be performed at randomization (Hour 0) and at 1, 2, 6, 24 hours after randomization, and on Day 5. Documentation of major adverse cardiac events (death, myocardial infarction, stroke, revascularization procedure with PCI or CABG)and serious adverse events (bleeding, other adverse events)will be performed until Day 5.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients with STEMI undergoing primary PCI with stenting
3. Informed consent obtained in writing

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Inability to give informed consent or high likelihood of being unavailable until the Day 5
* Prior PCI performed within 30 days prior to randomization
* Cardiogenic shock
* Major periprocedural complications (death, stent thrombosis, vessel perforation, arrhythmias requiring cardioversion, temporary pacemaker insertion or intravenous antiarrhythmic agents, respiratory failure requiring intubation, vascular injury (arteriovenous shunt, retroperitoneal bleeding), major bleeding (need for bood transfusion or drop in haemoglobin post-PCI by ≥ 5 gr/ dl or intracranial bleeding).
* Unsuccessful PCI (residual stenosis > 30% or flow < ΤΙΜΙ 3) or planned staged PCI in the next 5 days after randomization
* Requirement for oral anticoagulant prior to the Day 5 visit
* Current or planned therapy with other thienopyridine class of ADP receptor inhibitors.
* Known hypersensitivity to prasugrel or ticagrelor
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding.
* Any previous history of ischemic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
* Thombocytopenia (<100.000 / μL) at randomization
* Anaemia (Hct <30%) at randomization
* Polycytaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitors administration
* Severe allergy to contrast agent, unfractionated heparin, enoxaparin or bivalirudin that cannot be adequately premedicated.
* Recent (< 6 weeks) major surgery or trauma, including GABG.
* Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardiac events.
* Dialysis required.
* Severe uncontrolled chronic obstructive pulmonary disease
* Known severe hepatic impairement

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | 1hour
  Platelet reactivity Platelet assessed by VerifyNow P2Y12 assay 1 hour post randomization

SECONDARY OUTCOMES:
Platelet reactivity | 1 hour
  Platelet Reactivity assessed by Multiplate analyzer assay 1 hour post randomization
Platelet reactivity | 2 hours
  Platelet reactivity assessed by the VerifyNow assay 2 hours post randomization
Platelet reactivity | 2 hours
  Platelet Reactivity assessed by Multiplate analyzer 2 hours post randomization
Platelet reactivity | 6 hours
  Platelet Reactivity assessed by VerifyNow P2Y12 assay 6 hours post randomization
Platelet reactivity | 6 hours
  Platelet Reactivity assessed by Multiplate analyzer 6 hours post randomization
Platelet reactivity | 24 hours
  Platelet Reactivity assessed by VerifyNow P2Y12 assay 24 hours post randomization
Platelet reactivity | 24 hours
  Platelet Reactivity assessed by Multiplate analyzer 24 hours post randomization
Platelet reactivity | 5 days
  Platelet Reactivity assessed by VerifyNow P2Y12 assay 5 days post randomization
Platelet reactivity | 5 days
  Platelet Reactivity assessed by Multiplate analyzer 5 days post randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Patras University Hospital, Rio, Achaia, Greece

REFERENCES:
- [Derived] Alexopoulos D, Xanthopoulou I, Gkizas V, Kassimis G, Theodoropoulos KC, Makris G, Koutsogiannis N, Damelou A, Tsigkas G, Davlouros P, Hahalis G. Randomized assessment of ticagrelor versus prasugrel antiplatelet effects in patients with ST-segment-elevation myocardial infarction. Circ Cardiovasc Interv. 2012 Dec;5(6):797-804. doi: 10.1161/CIRCINTERVENTIONS.112.972323. Epub 2012 Nov 20. PMID 23169985